CLINICAL TRIAL: NCT04578509
Title: Evaluation of a Screening Program for SARS-CoV-2 Infection in the General Population Based on the Use of New Detection Approaches or for Diagnostic Orientation on Saliva (COVID-19)
Brief Title: Evaluation of a Screening Program for SARS-CoV-2 Infection in the General Population Based on the Use of New Detection Approaches or for Diagnostic Orientation on Saliva
Acronym: SALICOV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200960; 2020-A02431-38 (Other: APHP)
Record Dates: First submitted 2020-09-21; First posted 2020-10-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Screening program; SARS-CoV-2 infection
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva,axillary sweat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Salicov: Ambulatory adults or children requiring screening for SARS-CoV-2 by nasopharyngeal swab
  Interventions: Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: Saliva sample; Diagnostic Test: axillary sweat sample; Other: Data collection
- SalicovII (ancillary study): Ancillar study : Children and teachers / staff from middle and high schools in Ile de France Saliva samples is collected as part of care. Only a self-rated questionnaire is collected.
  Interventions: Diagnostic Test: Saliva sample; Other: Data collection

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — Research of SARS-CoV-2 infection in nasopharyngeal swab by RT-PCR and by antigenic test
  Groups: Salicov
Diagnostic Test: Saliva sample — Research of SARS-CoV-2 infection in saliva samples by RT-PCR and by new detection approach
Diagnostic Test: axillary sweat sample — Research of volatile olfactory compounds of SARS-CoV-2 infection by canine detection on axillary sweat.
  Groups: Salicov
Other: Data collection — Demographics, symptoms, medical history, acceptability of specimen, consumption in precedents hours are collected

SUMMARY:
The investigators hypothesize that detection of SARS-CoV2 on saliva samples will increase the performance of the screening program compared to the reference strategy (RT-PCR on a nasopharyngeal swab).

DETAILED DESCRIPTION:
Containment of the COVID19 pandemic relies on mass screening to allow rapid identification and isolation of cases to break transmission chains. The reference diagnostic method is based on detection of viral genomes by PCR on a nasopharyngeal swab sample (NPS).

However, the pandemic has generated a very high demand causing a shortage of specific swabs and difficulties in the supply of reagents and consumables. Nasopharyngeal sampling requires skilled personnel, and is sometimes poorly accepted by patients. These issues can reduce the quality of sampling and therefore the sensitivity of the test. This strategy also requires sending samples to specialized laboratories, generating a delay in providing results.

New diagnostic approaches on saliva samples are being developed allowing 1) an easier sampling procedure and 2) a diagnostic technique that can be performed in point-of-care.

Previous evaluations suggest that these approaches have a lower sensitivity than the reference strategy (PCR on NPS), around 50 to 90% depending on the technique used.

Despite lower sensitivity compared to the reference strategy, the investigators hypothesize that detection of SARS-CoV2 on saliva samples will improve the performance of the screening program by considerably increasing the number of individuals tested in shorter times.

The main objective of the study is to evaluate, for the detection of SARS-CoV-2 infection, the performance of various alternative virological diagnostic strategies on saliva samples, in comparison with the reference technique (RT-PCR on NPS).

The primary endpoint of the study is positivity of the standard technique (RT-PCR on NPS) for the SARS-CoV-2 virus. The result of the alternative strategies on a saliva sample will be considered as positive or negative according to criteria specific to each of them and compared to the result of the reference technique to estimate their respective sensitivity.

The secondary objectives are to compare the diagnostic performances of RT-PCR on saliva versus RT-PCR on NPS, the diagnostic performances of alternative techniques on saliva versus RT-PCR on saliva, to evaluate the acceptability of the saliva self-sampling and the cost-effectiveness of new diagnostic strategies compared to the reference technique.

The study will include adults and children in whom a NPS is performed for SARS-CoV-2 screening. After informed consent, participants will be asked to provide a saliva sample before nasopharyngeal sampling. Both samples will be analyzed in parallel. The analytical performance of each technique will be assessed, centrally or delocalised, depending on the feasibility of the techniques and according to the advice of the scientific board. The analyzes will be carried out by a team of technicians specifically recruited for the study. All samples collected will be stored in a centralized in a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child subject able to receive nasopharyngeal swab, regardless of age
* Subject in whom nasopharyngeal swab is performed for detection of SARS-CoV-2 as part of the screening system managed by APHP
* Subject or parent not opposed to saliva sampling and data collection as part of this research

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory adults or children requiring screening for SARS-CoV-2 by nasopharyngeal swab
Sampling Method: Probability Sample
Enrollment: 5197 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Positivity of RT-PCR on nasopharyngeal swab for the SARS-CoV-2 virus | At diagnosis
  RT-PCR on nasopharyngeal is considered as gold standard

SECONDARY OUTCOMES:
Positivity of RT-PCR on saliva sample for the SARS-CoV-2 virus | At diagnosis
Positivity of new detection approach on saliva sample for the SARS-CoV-2 virus | At diagnosis
Positivity of antigenic test on nasopharyngeal swab for the SARS-CoV-2 virus | At diagnosis
Practicability to samples | At diagnosis
  Number of samples tested in a day for each test
Practicability to premises | At diagnosis
  Quantity of premises required for each test
Practicability to interpretation | At diagnosis
  Feasibly Reading and interpretation For each test
Practicability to render time | At diagnosis
  Render times for each test
IgG Antibody detection in saliva | At diagnosis
  Research of IgG by ELISA and RDT
IgM Antibody detection in saliva | At diagnosis
  Research of IgM by ELISA and RDT
IgA Antibody detection in saliva | At diagnosis
  Research of IgA by ELISA and RDT
Positivity of canine olfactory detection of SARS-CoV-2 | At diagnosis
Patient tolerance of the salivary self-sampling | At diagnosis
  Evaluation by questionnaire of the patient tolerance of the salivary self-sampling compared to the nasopharyngeal swab (questions are about pain, discomfort, speed of performance)
Operator tolerance of the salivary self-sampling | At diagnosis
  Evaluation by questionnaire of the operator tolerance of the salivary self-sampling compared to the nasopharyngeal swab (questions is about pain, discomfort, speed of performance)
Cost of each approach | At diagnosis
  Including sampling, transport, technique (consumables, reagents, machine), human resources

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Le Goff, Professor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SARS-CoV-2 screening device of Assistance Publique des Hôpitaux de Paris (AP-HP), Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Lai CKC, Chen Z, Lui G, Ling L, Li T, Wong MCS, Ng RWY, Tso EYK, Ho T, Fung KSC, Ng ST, Wong BKC, Boon SS, Hui DSC, Chan PKS. Prospective Study Comparing Deep Throat Saliva With Other Respiratory Tract Specimens in the Diagnosis of Novel Coronavirus Disease 2019. J Infect Dis. 2020 Oct 13;222(10):1612-1619. doi: 10.1093/infdis/jiaa487. PMID 32738137
- [Background] Chen JH, Yip CC, Poon RW, Chan KH, Cheng VC, Hung IF, Chan JF, Yuen KY, To KK. Evaluating the use of posterior oropharyngeal saliva in a point-of-care assay for the detection of SARS-CoV-2. Emerg Microbes Infect. 2020 Dec;9(1):1356-1359. doi: 10.1080/22221751.2020.1775133. PMID 32459137
- [Background] Rao M, Rashid FA, Sabri FSAH, Jamil NN, Zain R, Hashim R, Amran F, Kok HT, Samad MAA, Ahmad N. Comparing Nasopharyngeal Swab and Early Morning Saliva for the Identification of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2021 May 4;72(9):e352-e356. doi: 10.1093/cid/ciaa1156. PMID 32761244
- [Background] Landry ML, Criscuolo J, Peaper DR. Challenges in use of saliva for detection of SARS CoV-2 RNA in symptomatic outpatients. J Clin Virol. 2020 Sep;130:104567. doi: 10.1016/j.jcv.2020.104567. Epub 2020 Jul 31. PMID 32750665
- [Background] Migueres M, Mengelle C, Dimeglio C, Didier A, Alvarez M, Delobel P, Mansuy JM, Izopet J. Saliva sampling for diagnosing SARS-CoV-2 infections in symptomatic patients and asymptomatic carriers. J Clin Virol. 2020 Sep;130:104580. doi: 10.1016/j.jcv.2020.104580. Epub 2020 Aug 5. No abstract available. PMID 32781366
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Background] Williams E, Bond K, Zhang B, Putland M, Williamson DA. Saliva as a Noninvasive Specimen for Detection of SARS-CoV-2. J Clin Microbiol. 2020 Jul 23;58(8):e00776-20. doi: 10.1128/JCM.00776-20. Print 2020 Jul 23. No abstract available. PMID 32317257
- [Background] McCormick-Baw C, Morgan K, Gaffney D, Cazares Y, Jaworski K, Byrd A, Molberg K, Cavuoti D. Saliva as an Alternate Specimen Source for Detection of SARS-CoV-2 in Symptomatic Patients Using Cepheid Xpert Xpress SARS-CoV-2. J Clin Microbiol. 2020 Jul 23;58(8):e01109-20. doi: 10.1128/JCM.01109-20. Print 2020 Jul 23. No abstract available. PMID 32414838
- [Background] Jamal AJ, Mozafarihashjin M, Coomes E, Powis J, Li AX, Paterson A, Anceva-Sami S, Barati S, Crowl G, Faheem A, Farooqi L, Khan S, Prost K, Poutanen S, Taylor M, Yip L, Zhong XZ, McGeer AJ, Mubareka S; Toronto Invasive Bacterial Diseases Network COVID-19 Investigators. Sensitivity of Nasopharyngeal Swabs and Saliva for the Detection of Severe Acute Respiratory Syndrome Coronavirus 2. Clin Infect Dis. 2021 Mar 15;72(6):1064-1066. doi: 10.1093/cid/ciaa848. PMID 32584972
- [Background] Lambert-Niclot S, Cuffel A, Le Pape S, Vauloup-Fellous C, Morand-Joubert L, Roque-Afonso AM, Le Goff J, Delaugerre C. Evaluation of a Rapid Diagnostic Assay for Detection of SARS-CoV-2 Antigen in Nasopharyngeal Swabs. J Clin Microbiol. 2020 Jul 23;58(8):e00977-20. doi: 10.1128/JCM.00977-20. Print 2020 Jul 23. No abstract available. PMID 32404480
- [Background] Azzi L, Baj A, Alberio T, Lualdi M, Veronesi G, Carcano G, Ageno W, Gambarini C, Maffioli L, Saverio SD, Gasperina DD, Genoni AP, Premi E, Donati S, Azzolini C, Grandi AM, Dentali F, Tangianu F, Sessa F, Maurino V, Tettamanti L, Siracusa C, Vigezzi A, Monti E, Iori V, Iovino D, Ietto G; ASST dei Sette Laghi Rapid Salivary Test Nurse staff Research Group; Grossi PA, Tagliabue A, Fasano M. Rapid Salivary Test suitable for a mass screening program to detect SARS-CoV-2: A diagnostic accuracy study. J Infect. 2020 Sep;81(3):e75-e78. doi: 10.1016/j.jinf.2020.06.042. Epub 2020 Jun 21. No abstract available. PMID 32579988
- [Background] Angle C, Waggoner LP, Ferrando A, Haney P, Passler T. Canine Detection of the Volatilome: A Review of Implications for Pathogen and Disease Detection. Front Vet Sci. 2016 Jun 24;3:47. doi: 10.3389/fvets.2016.00047. eCollection 2016. PMID 27446935
- [Background] Jendrny P, Schulz C, Twele F, Meller S, von Kockritz-Blickwede M, Osterhaus ADME, Ebbers J, Pilchova V, Pink I, Welte T, Manns MP, Fathi A, Ernst C, Addo MM, Schalke E, Volk HA. Scent dog identification of samples from COVID-19 patients - a pilot study. BMC Infect Dis. 2020 Jul 23;20(1):536. doi: 10.1186/s12879-020-05281-3. PMID 32703188
- [Background] Grandjean D, Sarkis R, Lecoq-Julien C, Benard A, Roger V, Levesque E, Bernes-Luciani E, Maestracci B, Morvan P, Gully E, Berceau-Falancourt D, Haufstater P, Herin G, Cabrera J, Muzzin Q, Gallet C, Bacque H, Broc JM, Thomas L, Lichaa A, Moujaes G, Saliba M, Kuhn A, Galey M, Berthail B, Lapeyre L, Capelli A, Renault S, Bachir K, Kovinger A, Comas E, Stainmesse A, Etienne E, Voeltzel S, Mansouri S, Berceau-Falancourt M, Dami A, Charlet L, Ruau E, Issa M, Grenet C, Billy C, Tourtier JP, Desquilbet L. Can the detection dog alert on COVID-19 positive persons by sniffing axillary sweat samples? A proof-of-concept study. PLoS One. 2020 Dec 10;15(12):e0243122. doi: 10.1371/journal.pone.0243122. eCollection 2020. PMID 33301539
- [Result] LeGoff J, Kerneis S, Elie C, Mercier-Delarue S, Gastli N, Choupeaux L, Fourgeaud J, Alby ML, Quentin P, Pavie J, Brazille P, Nere ML, Minier M, Gabassi A, Leroy C, Parfait B, Treluyer JM, Delaugerre C. Evaluation of a saliva molecular point of care for the detection of SARS-CoV-2 in ambulatory care. Sci Rep. 2021 Oct 26;11(1):21126. doi: 10.1038/s41598-021-00560-8. PMID 34702867
- [Result] Kerneis S, Elie C, Fourgeaud J, Choupeaux L, Delarue SM, Alby ML, Quentin P, Pavie J, Brazille P, Nere ML, Minier M, Gabassi A, Gibaud A, Gauthier S, Leroy C, Voirin-Mathieu E, Poyart C, Vidaud M, Parfait B, Delaugerre C, Treluyer JM, LeGoff J. Accuracy of saliva and nasopharyngeal sampling for detection of SARS-CoV-2 in community screening: a multicentric cohort study. Eur J Clin Microbiol Infect Dis. 2021 Nov;40(11):2379-2388. doi: 10.1007/s10096-021-04327-x. Epub 2021 Aug 3. PMID 34342768